CLINICAL TRIAL: NCT03257371
Title: A Biologic Joint Replacement Strategy to Treat Patients With Severe Knee Trauma and Post-Traumatic Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: James Stannard (Other)
Responsible Party: Sponsor-Investigator, James Stannard, Chairman, Department of Orthopaedic Sugery; Medical Director, Missouri Orthopaedic Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Other Study IDs: 2002751
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Post-traumatic Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-traumatic knee OA: post-traumatic knee OA and requiring a tibial plateau and meniscus arthroplasty plus a femoral condyle arthroplasty

SUMMARY:
With IRB approval and informed consent, patients (n=10) (18-50 years old) with post-traumatic knee OA and requiring a tibial plateau and meniscus arthroplasty plus a femoral condyle arthroplasty will be enrolled in the study. Primary criteria for inclusion will be Grade IV changes in the articular cartilage of the femoral condyle and tibial plateau and meniscal pathology in the medial or lateral femorotibial joint as determined by physical examination, diagnostic imaging and knee arthroscopy by the PI. Exclusion criteria include Grade III or IV changes in any other compartment of the knee, acute injury to any other part of the affected lower extremity, or inability to comply with the protocol.

After enrollment, patients will undergo standardized knee radiography, and complete assessments (described below). Size-matched (standard clinical methodology) proximal tibia with meniscus and distal femur allografts from the same donor will be obtained from a tissue bank (Musculoskeletal Transplant Foundation, Edison, NJ) who has licensed the MOPS technology. The medial or lateral femoral condyle will be replaced using our novel instrumentation and technique described above. Tibial plateau-meniscus grafts will be trimmed and used to replace the entire medial or lateral tibial condyle while sparing the attachments of ACL, PCL and respective collateral ligament. The tibial plateau graft will be fixated using commercial available implants used for bone fixation. In the event that the meniscus has been detached from the tibial plateau during graft harvest, the periphery of the meniscus will be sutured to the capsule following standard meniscus transplant procedure.

Patients will undergo controlled post-operative rehabilitation according to standard protocols for osteochondral with concurrent meniscus allografts.

Range of motion, VAS pain score, SF-12, Tegner score, International Knee Documentation Committee (IKDC) subjective and objective scores, PROMIS Bank v1.2 - Physical Function-Mobility, PROMIS v1.1 - Global Health, PROMIS Bank v1.1- Pain Interference, PROMIS Bank v1.2 - Physical Function and Marx score as well as complete radiographs of the affected knee will be obtained prior to surgery and at 6 weeks, 3 months, 6 months, and 12 months after surgery to evaluate healing, function and evidence for arthrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring repair via tibial plateau and meniscus arthroplasty plus a femoral condyle arthroplasty
2. The subject is able and willing to consent to participate in the study

Exclusion Criteria:

1. Acute injury to any other part of the affected lower extremity
2. The subject is unwilling, or unable to consent due to psychiatric condition or legal incompetence
3. BMI > 40
4. Age > 50 at the time of enrollment
5. The subject is either pregnant, or a prisoner
6. Currently involved in a workers' compensation case at the time of enrollment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients (n=10) (18-50 years old) with post-traumatic knee OA and requiring a tibial plateau and meniscus arthroplasty plus a femoral condyle arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Stannard, MD, Principal Investigator — University of Missouri, Department of Orthopaedic Surgery
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-traumatic Knee OA
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: This study was fully enrolled.
Arm/Group | Post-traumatic Knee OA
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.4 [34 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale Pain Score
Description: patient reported Visual Analogue Scale Pain Score, 0 no pain, 10 maximum pain
Time Frame: 12 months
Population: 7 patients completed the study without needing revision/TKA surgery or being lost to follow-up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Post-traumatic Knee OA
Number analyzed (Participants) | 7
units on a scale | 2.3 [0 to 7]

2. Secondary Outcome: Tegner Activity Level Scale
Description: Patient reported outcome scale related to work and sporting activities, The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Time Frame: 12 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Post-traumatic Knee OA
Number analyzed (Participants) | 7
units on a scale | 3.3 [2 to 4]

3. Secondary Outcome: International Knee Documentation Committee (IKDC) Total Score
Description: Knee specific patient reported outcome, ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Time Frame: 12 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Post-traumatic Knee OA
Number analyzed (Participants) | 7
units on a scale | 50.6 [39.1 to 64.4]

4. Secondary Outcome: PROMIS - Physical Function and Mobility
Description: A survey related to physical function and mobility, T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric:
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. A higher score is better for this outcome measure as it indicates more function/mobility compared to the mean of the reference population.
Time Frame: 12 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Post-traumatic Knee OA
Number analyzed (Participants) | 7
units on a scale
  Physical Function | 41.2 [27.7 to 46.6]
  Mobility | 43.1 [37.7 to 47.9]

ADVERSE EVENTS:
Time Frame: AE data was followed for one year.
Description: AE:
  I. Bleeding II. Infection III. Pain that is uncontrolled with standard post-operative analgesia protocol
  SAE:
  I. Bleeding that is significant enough to require extended hospitalization or unplanned critical care interventions II. Infection that is significant enough to require extended hospitalization or unplanned critical care interventions III. Pain that is significant enough to require extended hospitalization or unplanned critical care interventions
Arm/Group | Post-traumatic Knee OA
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-traumatic Knee OA (N=10)
Revision or TKA surgery (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-traumatic Knee OA (N=10)
Bone Grafting (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee Arthroscopy (Musculoskeletal and connective tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
1 Patient was lost to follow-up after their 6 week follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT03257371/Prot_SAP_000.pdf